CLINICAL TRIAL: NCT04607538
Title: The Faroese Knee Cohort: An Investigation of Etiology and Long-term Implications of Trochlear Dysplasia and Patellar Dislocations
Brief Title: The Faroese Knee Cohort: Etiology and Long-term Implications of Trochlear Dysplasia and Patellar Dislocations.
Acronym: FKC
Status: Recruiting | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristoffer Barfod, MD. Ph.D. Associate Professor, Hvidovre University Hospital
Other Study IDs: FaroeseKneeCohort
Record Dates: First submitted 2020-06-18; First posted 2020-10-29 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Patellar Dislocation; ACL Injury; Meniscus Lesion; Trochlear Dysplasia
Keywords: Patellar instability; Patellar dislocation; ACL-rupture; Meniscus lesion; Meniscus injury
MeSH Terms: conditions — Patellar Dislocation; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patellar dislocation, but no trochlear dysplasia: This group consist of patients in age from 15-20 years old in the Faroe Islands, who experience patellar dislocation, but do not have femoral trochlear dysplasia measured on MRI or X-ray
  Interventions: Other: No intervention is made
- Patiens with patellar dislocation and trochlear dysplasia: This group consists of patients in the age from 15-20 years old in the Faroe Islands, who have experience one or more patellar dislocations and have femoral trochlear dysplasia measured on MRI or X-ray
  Interventions: Other: No intervention is made
- Patients with other knee injury: This group consists of patients in the age from 15-20 years old in the Faroe Islands, who have had an ACL-rupture or an meniscus injury.
  Interventions: Other: No intervention is made

INTERVENTIONS:
Other: No intervention is made — No intervention is made. This i an observational study.

SUMMARY:
The investigators intend to establish a national cohort including all persons in the ages from 15-20 years old with patellar instability (PI) or a prior knee injury (ACL-ruptur or meniscus damage) . The cohort will be nicknamed "The Faroese Knee Cohort".

The overall aim is to investigate two groups.

1. The patella instability group, in which we intend to investigate the following.

   * Prevalence of patellar dislocation and trochlear dysplasia in the Faroe Islands.
   * Risk factors for patellar dislocations-
   * Heredity of trochlear dysplasia.
   * If there is a specific gene responsible for the development of trochlear dysplasia.
   * The development of retropatellar artrhosis, its onset and its impact on quality of life and function,
2. Knee injury group (ACL-ruptur or meniscus injury)

   * The prevalence of ACL-rupture and/or meniscus injury in this specific group in the Faroe Islands.
   * The impact on quality of life and function.

DETAILED DESCRIPTION:
The Faroese Knee Cohort aims to consist of all persons in the Faroe Island between 15-20 years old with patellar instability* (PI) or a knee injury.

Special focus will be on PI, Patella dislocation (PD) and Trochlear Dysplasia (TD), a condition where the femoral trochlea has a dysplastic shape and lacks the lateral support of the patella. The diagnosis will be set by MRI of the knees and is in this study defined as the presence of one of the following: Crossing sign on a true lateral x-ray, lateral trochlear inclination angle < 11 degrees or a trochlear depth < 3 mm.

The hypothesis is that abnormal values in the following measures will be associated with increased risk of patellar dislocation and worse patient reported outcome: Caton-Deschamps index, Lateral Trochlear Inclination, Trochlear Facet Asymmetry, Trochlear Depth, Tuberostias Tibia - Trochlear Groove distance, Patello-trochlear index and Tuberositas Tibia - Posterior Cruciate Ligament distance.

Furthermore, we expect pivoting sports to be a behavioral risk factor.

The primary endpoint is measured by the number of patellar dislocations or near-dislocation the patient experiences (daily, weekly, monthly, yearly).

The secondary endpoint is the patient reported outcome measures.

*Definition: Patellar instability (PI) is the overall term encompassing both 1) recurrent patella dislocations and 2) recurrent episodes of a clear sensation of the kneecap riding on the outer border/aspect of the knee before popping back in track. The episodes must be a severe complaint for the patient. PI usually follows after a first time patellar dislocation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15-20 years at the start of patient enrolment.
* The feeling of patellar instability, or patellar dislocation/near-dislocation.
* The person has to be from the Faroe Islands.
* All persons under the age of 18 must get written consent by their parents

Exclusion Criteria:

* Terminal illness
* Mental disabilities and illness, meaning that the patient cannot independently answer the PROM´s and cooperate to the clinical investigation.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients must either live or be born in the Faroe Islands, as this is a national cohort study. They will be invited to join the study if the live up to the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2051-12-01 (Estimated)

PRIMARY OUTCOMES:
Severity of patellar dislocations | 1 year
  The severity of PD defined by number of PD or near-dislocations the patient experience (daily, weekly, monthly, yearly).

SECONDARY OUTCOMES:
Risk factors for patellar dislocation 1 | 1 year
  The investigators will investigate if there is an correlation between the amount of patellar dislocations and the following measurements Caton-Deschamps index: Measuring in the ratio from 0-2. (normal 0.6-1.3, patella alta: > 1.3, Patella Baja: <0,6)
Risk factors for patellar dislocation 2 | 1 year
  The investigators will investigate if there is an correlation between the amount of patellar dislocations and the following measurements:
  Lateral Trochlear Inclination: Measured in degrees, the range from 0-20 degrees. (< 11 degrees indicates trochlear dysplasia)
Risk factors for patellar dislocation 3 | 1 year
  The investigators will investigate if there is an correlation between the amount of patellar dislocations and the following measurements:
  Trochlear Facet Asymmetry: Measured in the ratio from 0-1. ( < 0.4 indicates trochlear dysplasia)
Risk factors for patellar dislocation 4 | 1 year
  The investigators will investigate if there is an correlation between the amount of patellar dislocations and the following measurements:
  Trochlear Depth: Measured in centimeters in the range from 0-3 cm. (< 3 cm is abnormal)
Risk factors for patellar dislocation 5 | 1 year
  The investigators will investigate if there is an correlation between the amount of patellar dislocations and the following measurements:
  Tuberositas Tibia - Trochlear Groove distance': Measured in mm, in the range from 0-25 mm (< 15 mm is normal, 15-20 is borderline, > 20 mm is abnormal)
Risk factors for patellar dislocation 6 | 1 year
  The investigators will investigate if there is an correlation between the amount of patellar dislocations and the following measurements:
  Patello-trochlear index: Is measured in a ratio in percentages. Measurements from 0-100%. (Normal range: 0.18-0.80, patella alta < 0.18, patella baja >0.80)
Patient reported activity | 1 year
  The patient reported outcome measured by the following measurements:
  MARX score (Activity score),
Patient reported luxation score | 1 year
  The patient reported outcome measured by the following measurements
  - Banff Patella Instability Instrument (Luxation score)
Patient reported patellofemoral pain | 1 year
  The patient reported outcome measured by the following measurements
  * The Kujala score (Patellofemoral pain score)

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No